CLINICAL TRIAL: NCT04729166
Title: Effectiveness of Structured Education and Follow-up on Management of Perceived Breastmilk Insufficiency: A Randomized Control Trial
Brief Title: The Management of Perceived Breastmilk Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Zekiye Karaçam, Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Interventional
Record Dates: First submitted 2021-01-16; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Breast Milk Expression; Breast Feeding, Exclusive
Keywords: breastmilk; breastfeeding; education; follow-up
MeSH Terms: conditions — Breast Milk Expression; Breast Feeding

STUDY DESIGN:
Intervention Model Description: Following recruitment, the pregnant women were divided into a study and a control group by randomization (1:1 randomization)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The study group were provided with education with structured educational material and followed in this study, in addition to the usual care provided by healthcare professionals.
  Interventions: Behavioral: Structured education and follow-up
- Control group (No Intervention): Control group was int the usual care.

INTERVENTIONS:
Behavioral: Structured education and follow-up — This structured educational material was developed by the authors on the basis of the literature. Interventions of the study were carried out in the 32nd-42nd week of pregnancy, 3rd-7th day postpartum, and at the 1st month. At first stage, a 15-20-minute education was given to the pregnant women in the study group in the breastfeeding room of the facility, educational booklets were distributed. The main emphasis parts of the education were repeated with a standard summary information form at each follow-up.
  Arms: Study group

SUMMARY:
A randomized control trial was made to determine the effectiveness of structured education and follow-up in the management of perceived milk insufficiency among breastfeeding mothers.

DETAILED DESCRIPTION:
Mothers 'perception of breastmilk insufficiency are important conditions affecting babies' exclusively breastfeeding in the first six months.

This study was made to determine the effectiveness of structured education and follow-up in the management of perceived breastmilk insufficiency among breastfeeding mothers. It was tested the hypotheses that there are no differences between mothers who have been provided with structured education and follow-up and those who have not received the education in terms of initiating breastfeeding in the first one hour, breastmilk insufficiency perceptions, the rate of exclusive feeding of breast milk to babies 0-2 months old, the baby's amount of milk intake and weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Women in their 32nd-42nd week of pregnancy
* Being literate in Turkish
* Being at least a primary school graduate

Exclusion Criteria:

* Having a history of psychological or mental health problems
* Having any condition in the mother or infant that was a barrier to breastfeeding
* The baby's admission into the neonatal unit
* The baby's separation from the mother for any reason

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 70 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
The starting breastfeeding in the first hour | Postpartum 3rd-7th day
  assessed using the Breastfeeding Follow-up Form in 3rd-7th day postpartum. Mothers reported whether they started breastfeeding within the first hour after birth.
Bottle-feeding | Postpartum 3rd-7th day
  assessed using the Breastfeeding Follow-up Form in 3rd-7th day postpartum. Mothers reported whether they feed her baby with bottle-feeding.
The baby's amount of milk intake | Postpartum 3rd-7th day
  assessed using The Scoring System for Measuring a Baby's Intake of Breast Milk. This measurement tool was developed to assess the amount of breast milk a baby is fed. The form is made up of 5 sections: the baby's weight, state of satisfaction, frequency and characteristics of urination and defecation and the condition of the mother's breasts. This tool is filled by observation, measurement and interview. The tool rates each status on the basis of 0, 1 or 2, the highest possible total score being 10. A score of 8-10 indicates that the intake of breast milk is good, 0-7 indicates an insufficient intake.
The baby's amount of milk intake | Postpartum the 1st month
  assessed using The Scoring System for Measuring a Baby's Intake of Breast Milk. This measurement tool was developed to assess the amount of breast milk a baby is fed. The form is made up of 5 sections: the baby's weight, state of satisfaction, frequency and characteristics of urination and defecation and the condition of the mother's breasts. This tool is filled by observation, measurement and interview. The tool rates each status on the basis of 0, 1 or 2, the highest possible total score being 10. A score of 8-10 indicates that the intake of breast milk is good, 0-7 indicates an insufficient intake.
The baby's amount of milk intake | Postpartum 2nd month
  assessed using The Scoring System for Measuring a Baby's Intake of Breast Milk. This measurement tool was developed to assess the amount of breast milk a baby is fed. The form is made up of 5 sections: the baby's weight, state of satisfaction, frequency and characteristics of urination and defecation and the condition of the mother's breasts. This tool is filled by observation, measurement and interview. The tool rates each status on the basis of 0, 1 or 2, the highest possible total score being 10. A score of 8-10 indicates that the intake of breast milk is good, 0-7 indicates an insufficient intake.
Exclusively feeding with mother's milk | Postpartum 3rd-7th day
  assessed using the Breastfeeding Follow-up Form. Mothers reported whether they feed her baby with exclusively mother's milk.
Exclusively feeding with mother's milk | Postpartum the 1st month
  assessed using the Breastfeeding Follow-up Form. Mothers reported whether they feed her baby with exclusively mother's milk.
Exclusively feeding with mother's milk | Postpartum 2nd month
  assessed using the Breastfeeding Follow-up Form. Mothers reported whether they feed her baby with exclusively mother's milk.
Believing breast milk is adequate | Postpartum 3rd-7th day
  assessed using the Breastfeeding Follow-up Form. Mothers reported whether they believed her baby take adequate breast milk.
Believing breast milk is adequate | Postpartum the 1st month
  assessed using the Breastfeeding Follow-up Form. Mothers reported whether they believed her baby take adequate breast milk.
Believing breast milk is adequate | Postpartum 2nd month
  assessed using the Breastfeeding Follow-up Form. Mothers reported whether they believed her baby take adequate breast milk.

SECONDARY OUTCOMES:
Baby's height | Postpartum 3rd-7th day
  used to determine the baby's height. Baby's height was measured and recorded by the researcher to The Breastfeeding Follow-up Form as cm.
Baby's height | Postpartum 1st month
  used to determine the baby's height. Baby's height was measured and recorded by the researcher to The Breastfeeding Follow-up Form as cm.
Baby's height | Postpartum 2nd month
  used to determine the baby's height. Baby's height was measured and recorded by the researcher to The Breastfeeding Follow-up Form as cm.
Believing the baby is adequately fed. | Postpartum 3rd-7th day
  assessed using the Breastfeeding Follow-up Form. Mothers reported whether they believed her baby fed adequate.
Believing the baby is adequately fed. | Postpartum 1st month
  assessed using the Breastfeeding Follow-up Form. Mothers reported whether they believed her baby fed adequate.
Believing the baby is adequately fed. | Postpartum 2nd month
  assessed using the Breastfeeding Follow-up Form. Mothers reported whether they believed her baby fed adequate.
Being satisfied with baby's weight gain. | Postpartum 3rd-7th day
  assessed using the Breastfeeding Follow-up Form. Mothers reported whether they were satisfied from her baby's weight gain.
Being satisfied with baby's weight gain. | Postpartum 1st month
  assessed using the Breastfeeding Follow-up Form. Mothers reported whether they were satisfied from her baby's weight gain.
Being satisfied with baby's weight gain. | Postpartum 2nd month
  assessed using the Breastfeeding Follow-up Form. Mothers reported whether they were satisfied from her baby's weight gain.
Baby's weight | Postpartum 3rd-7th day
  used to determine the baby's weight. Baby's weight was measured and recorded by the researcher to The Breastfeeding Follow-up Form as grams.
Baby's weight | Postpartum 1st month
  used to determine the baby's weight. Baby's weight was measured and recorded by the researcher to The Breastfeeding Follow-up Form as grams.
Baby's weight | Postpartum 2nd month
  used to determine the baby's weight. Baby's weight was measured and recorded by the researcher to The Breastfeeding Follow-up Form as grams.

CONTACTS AND LOCATIONS:
Overall Officials: Zekiye Karaçam, Prof. Dr., Study Chair — Adnan Menderes University, Faculty of Health Sciences, Division of Midwifery
Locations (1):
- Aydın Adnan Menderes University, Faculty of Health Sciences, Division of Midwifery, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.